CLINICAL TRIAL: NCT00338325
Title: A Randomized Trial Of Reading Preoperatively To Day Surgery Children To Reduce Anxiety and Pain
Brief Title: Reading Preoperatively to Reduce Anxiety in Day Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: IWK Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3317; IWK studentship award
Record Dates: First submitted 2006-06-15; First posted 2006-06-20 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Pre-operative Pediatric Anxiety
Keywords: Pediatric Anxiety; Pediatric Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment (Experimental): 50% randomized to receive treatment: reading pre-operatively
  Interventions: Behavioral: Reading program
- Control (No Intervention): 50% randomized to receive no intervention pre-operatively: no reading

INTERVENTIONS:
Behavioral: Reading program — Reading of children's story/picture books preoperatively
  Arms: Treatment

SUMMARY:
This study is designed to implement the reading of age appropriate books by a trained reader into the waiting area of a pediatric day surgery unit to determine if it is effective at reducing the anxiety and pain levels of parents and children by providing a safe and calming activity for the child. This is a single-centre trial based at the IWK Health Centre. The primary outcome will be based on the anxiety and pain scores of the research participants.

DETAILED DESCRIPTION:
The purpose of this study is 1. to investigate the child and parental anxiolytic effects of reading age-appropriate books by Read To Me readers to the children in the waiting room of day surgery units 2. to investigate if parents use reading to assist their children during their recovery period at home and the impact of this effort. Participants will be asked to report their feelings of anxiety before and after being read to using Kuttner's face scale of anxiety and Speilberger's State-Trait Anxiety Inventory (STAI) for the adults. If the child is less than 5 years of age, a proxy measure of child anxiety will be taken. The anxiety measures will be taken immediately after consent is obtained and then will be taken again 20-60 minutes later. The exact time the second measure is taken after initial anxiety measurements will be recorded. This procedure will be used for both experimental and control groups. Parents will also be asked to fill out Conners' Parent Rating Scale - Revised to assess the usual temperament of their child. Parents and children will be approached to participate in the present study. Consent to be read to and consent to participate in the study will be separated. Families may consent to be read to without consenting to the research. As is the routine in other areas of the hospital, parents will be verbally asked for consent to read to their children by the Read To Me staff. Two trained readers from the Read To Me program at the IWK Health Centre will provide the reading of age-appropriate books to participants in the experimental group.

Research personnel will obtain written consent for participation in the research. The Read To Me activities will include being read to and receiving an activity bag with an age-appropriate paper back book chosen by experienced literacy practitioners, a related craft and literacy activity the child can complete at home after reading the story and a brochure for parents which lists age-specific literacy skills, recommended book lists and reading tips which explain how to share books with children.

Parents will then be asked a few questions in a semi structured qualitative interview regarding their experience in the waiting room. Two days after surgery a follow up interview will take place on the telephone that will include information the parents recorded in the diary they were given at the time of participation in the study. Parents will be given the diary at the time of consent where the child's pain with activity (2-3 times daily), the child's anxiety (2-3 times daily) and the use of distracters during recovery can all be recorded.

Two hundred and fifty two day surgery patients and their parents were assessed for eligibility. 52 refused to participate and 2 parents withdrew from the study because they were not interested in continuing with the research. Two hundred children and their parents were recruited for participation and were randomly assigned by cluster determined by the day they came to surgery to either the control or the experimental group. One hundred and eighteen participants were allocated to the experimental group while eighty-two participants were allocated to the control group.

Both groups will be evaluated for outcome results and will be compared to determine if there is a difference in the anxiety and pain scores collected for each group. It is expected that the children who were in the reading group will report less anxiety and pain during day surgery and during recovery than the children who received usual care.

ELIGIBILITY:
Inclusion Criteria:

* 2-8 years old and their parents
* who are undergoing Day Surgery at the IWK Health Centre will be eligible to participate in this study.

Exclusion Criteria:

* children of parents who have not consented to participation in the study will be ineligible to participate.
* Any parent or child not having a signed authorization form will be ineligible to participate.

Ages: 2 Years to 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 200 (Actual)
Dates: Start 2005-06; Primary Completion 2005-06 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Kuttner's face scale of anxiety for children | pre & post surgery
Speilberger's State-Trait Anxiety Inventory (STAI) for the adults. | pre & post

SECONDARY OUTCOMES:
Conners' Parent Rating Scale - Revised - Hyperactive and Anxiety scores | pre
Data from Semi-Structured Qualitative Parental Interviews | post surgery

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J. McGrath, PhD., Principal Investigator — IWK Health Centre